CLINICAL TRIAL: NCT07061873
Title: Physical Exercise Program for Adults With Diffuse Interstitial Lung Disease in a Pulmonary Rehabilitation Context
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de La Frontera (Other)
Responsible Party: Principal Investigator, Sayen Huaiquilaf-Jorquera, Physical Therapist; Specialist in Ventilatory Terapy; Master in Innovation of Universitary Pedagogy in Education Science; Academic Department Science of Rehabilitation, University of La Frontera, Universidad de La Frontera
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECA RP-EPID; DI24-011 (Other Grant/Funding Number: Universidad de La Frontera)
Record Dates: First submitted 2025-03-21; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Interstitial Lung Disease Due to Systemic Disease (Disorder); Interstitial Lung Disease in Patients With Rheumatoid Arthritis; Pulmonary Fibrosis
Keywords: ILD; Pulmonary rehabilitation; aerobic excercise; limb strenght; respiratory muscle strenght
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Other): Control (Aerobic excercise)
  Interventions: Procedure: Aerobic excersise
- Intervention (Experimental): Intervention (Muscle strength limbs, inspiratory muscle strength, aerobic exercise)
  Interventions: Procedure: Aerobic excersise; Procedure: Muscle strength limbs, inspiratory muscle strength

INTERVENTIONS:
Procedure: Aerobic excersise — 20 aerobic exercise sessions, with a duration of 45 to 60 minutes, for 10 weeks.
Procedure: Muscle strength limbs, inspiratory muscle strength — 20 sessions of exercise Muscle strength limbs, inspiratory muscle strength, with a duration of 60 minutes, for 10 weeks
  Arms: Intervention

SUMMARY:
This study aims to evaluate the effectiveness of an exercise program that includes three exercise modalities (Aerobic, Limb Strength and Respiratory Muscle Strength) versus an exercise program that includes only one modality (Aerobic) in the context of a Pulmonary Rehabilitation program in adults with diffuse interstitial disease in the Araucanía Region, in terms of exercise tolerance.

A randomized clinical trial will be conducted, with 2 parallel groups, with masked evaluator. This study will include adults with a diagnosis of Diffuse Interstitial Lung Disease who are referred according to their medical condition and who agree to participate through an informed consent form. Participants will be recruited in the community and will be referred to the Physical Function and Rehabilitation Laboratory of the Faculty of Medicine of the Universidad de La Frontera, where they will be evaluated and subsequently randomly assigned to each group. The evaluation consists of a series of tests and instruments to collect information regarding dyspnea, exercise tolerance, muscle strength and lung function, among others. The intervention corresponds to a Pulmonary Rehabilitation program, where both groups will receive education in psychological and nutritional aspects, self-care and physical activity. The difference between groups is that the control group will receive an intervention with an aerobic exercise modality and the experimental group will receive three exercise modalities together (aerobic, strengthening of extremities and strengthening of respiratory muscles).The program will last 10 weeks, with sessions twice a week, and at the end of the program the initial parameters will be re-evaluated.

Data analysis will be performed using descriptive statistical elements, such as distribution tables and graphs. The inferential analysis will be performed using Chi2 for the association between the intervention and the main outcome variable, in addition to the calculation of RR to assess the magnitude of the association; the secondary outcome variables will be calculated for the primary outcome variable association; secondary outcome variables will be analyzed using Student's t-test.

DETAILED DESCRIPTION:
General Objective: To evaluate the effectiveness of an exercise program that includes three exercise modalities (Aerobic, Limb Strength and Respiratory Muscle Strength) versus an exercise program that includes only one modality (Aerobic) in the context of a Pulmonary Rehabilitation program in adults carriers of diffuse interstitial disease in the Araucanía Region, in terms of exercise tolerance.

Specific Objectives:

1. To evaluate the effectiveness of an exercise program that includes three modalities (Aerobic, Limb Strength and Respiratory Muscle Strength) versus an exercise program of only one modality (Aerobic) in the context of a Pulmonary Rehabilitation program in adults carriers of diffuse interstitial disease in the Araucanía Region, in terms of exercise tolerance.
2. To evaluate the effectiveness of an exercise program with three modalities (Aerobic, Limb Strength and Respiratory Muscle Strength) versus a one-modality exercise program (Aerobic) within a Pulmonary Rehabilitation program in adults with diffuse interstitial disease in the Araucanía Region, in terms of dyspnea control.
3. To evaluate the effectiveness of an exercise program with three modalities (Aerobic, Limb Strength and Respiratory Muscle Strength) versus an exercise program with one modality (Aerobic) within a Pulmonary Rehabilitation program in adults with diffuse interstitial disease in the Araucanía Region, in Health-Related Quality of Life.
4. To evaluate the effectiveness of an exercise program with three modalities (Aerobic, Limb Strength and Respiratory Muscle Strength) versus an exercise program with one modality (Aerobic) within a Pulmonary Rehabilitation program in adults with diffuse interstitial disease of the Araucanía Region, in terms of upper limb strength.
5. To evaluate the effectiveness of an exercise program with three modalities (Aerobic, Limb Strength and Respiratory Muscle Strength) versus an exercise program with one modality (Aerobic) within a Pulmonary Rehabilitation program in adults with diffuse interstitial disease in the Araucanía Region, in terms of lower limb strength.
6. To evaluate the effectiveness of an exercise program with three modalities (Aerobic, Limb Strength and Respiratory Muscle Strength) versus an exercise program with one modality (Aerobic) within a Pulmonary Rehabilitation program in adults with diffuse interstitial disease in the Araucanía Region, in terms of inspiratory muscle strength.
7. To evaluate the effectiveness of an exercise program with three modalities (Aerobic, Limb Strength and Respiratory Muscle Strength) versus an exercise program with one modality (Aerobic) within a Pulmonary Rehabilitation program in adults with diffuse interstitial disease in the Araucanía Region, in pulmonary function.
8. To evaluate the adherence to treatment of an exercise program with three modalities (Aerobic, Limb Strength and Respiratory Muscle Strength) and the exercise program of one modality (Aerobic) in the context of a Pulmonary Rehabilitation program in adults with diffuse interstitial disease in the Araucanía Region.
9. To evaluate the incidence of adverse effects that lead to stopping the exercise session according to the exercise program: with three modalities (Aerobic, Limb Strength and Respiratory Muscle Strength) versus a one-modality exercise program (Aerobic) in the context of a Pulmonary Rehabilitation program in adults with diffuse interstitial disease in the Araucanía Region.
10. To describe the functionality in users who enter the Pulmonary Rehabilitation program for adults with diffuse interstitial disease in the Araucanía Region.
11. To describe the cognitive function in users who enter the Pulmonary Rehabilitation program for adults with diffuse interstitial disease in the Araucanía Region.

Design It corresponds to a randomized clinical trial, 2 parallel groups, with masked evaluator. This design is the one that provides the best certainty of evidence to attribute causality, therefore, to evaluate the effectiveness of an intervention.

Sample The study population will be adults with a medical diagnosis of diffuse lung disease, clinically stable, who are under medical treatment (In the original text it said: "in the Polyclinic of Respiratory Diseases", however, due to the sample size obtained, as a team we decided to make a free invitation to those who wish to participate and are under medical treatment in the public or private sector).

The sample will be constituted by participants who meet the following eligibility criteria:

Inclusion Criteria.

* Adults aged 18 years or older.
* Medical diagnosis of diffuse interstitial lung disease.
* Medical referral to pulmonary rehabilitation according to stability criteria.
* Signing of the Informed Consent form.

Exclusion Criteria

* Neuromotor impairment that prevents independent transfer.
* Cognitive deficit preventing him/her from understanding simple instructions.
* General contraindications to exercise according to the American College of Sports Medicine.

In the sample size calculation, a number of 26 subjects was obtained, considering a significance level of 5%, a power of 80%, an estimated difference between the groups under study of 40 (±35) meters walked in the main response variable, evaluated with the 6-minute Walk Test (De las Heras JC, Hilberg O, Lokke A, Bendstrup E. Tele-rehabilitation program in Idiopathic Pulmonary Fibrosis. European Respiratory Journal. 2019). Considering a 10% loss, the final sample size will be 29 individuals.

Evaluation: A set of physical assessments and questionnaires that evaluate the following.

functional parameters:

* Exercise tolerance
* Dyspnea
* Health-Related Quality of Life
* Limb Muscular Strength
* Respiratory Muscular Strength
* Pulmonary Function
* Functionality
* Cognition

Training: is the intervention itself and consists of aerobic physical exercise or a combination of 3 modalities:

* Aerobic Exercise
* Limb Strength Exercise
* Respiratory Muscular Strength Exercise

All interventions will take place at the Faculty of Medicine of the Universidad de La Frontera, located at Claro Solar 115, and the Laboratory of Physical Fitness and Rehabilitation of the Universidad de La Frontera, located at 18 de Septiembre 525, 6th floor.

This research has been approved by the Scientific Ethics Committee of Universidad de La Frontera, Act Number 119_2024.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older.
* Medical Diagnosis of Diffuse Interstitial Pulmonary Disease.
* Medical Referral to pulmonary rehabilitation according to stability criteria.
* Sign the Informed Consent form.

Exclusion Criteria:

* Neuromotor impairment that prevents independent transfer.
* Cognitive deficit that prevents you from understanding simple instructions.
* General exercise contraindications according to the American College of Sports Medicine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Exercise tolerance | Baseline and then at the end of the 10-week training period
  It is the body's ability to withstand physical activity. It is measured by the duration and intensity of exercise that a person can perform without excessive fatigue, pain or shortness of breath.

SECONDARY OUTCOMES:
Perceived effort | Baseline and then at the end of the 10-week training period
  Corresponds to the subjective feeling of how demanding a physical activity is. It reflects the intensity with which one feels one's body is working, from "very light" to "maximum effort". It is a useful tool for regulating exercise intensity according to the patient's perception. For the purposes of this study, the perception of exertion will be assessed using the Modified Borg Scale from 0 to 10 points, where 0 corresponds to "No dyspnea" and 10 "Very, very severe".
Dyspnea | Baseline and then at the end of the 10-week training period
  Subjective sensation of shortness of breath or difficulty breathing. It may be mild or severe, acute or chronic. It is a frequent symptom of various pulmonary or cardiac conditions, but may also be due to anxiety or intense exercise. To assess Dyspnea, we use the Modified Medical Research Council (mMRC) scale, where 0 is "No shortness of breath except during strenuous exercise" and 4 is "Choking sensation during day-to-day exertion such as getting dressed or going out of the house and need for rest".
Inspiratory muscle strength | Baseline and then at the end of the 10-week training period
  Inspiratory muscle strength is the ability of the respiratory muscles to expand the lungs during inspiration. It is measured by the maximum pressure they can generate when breathing in against resistance. A good level of inspiratory strength is crucial for efficient breathing and good lung health. It will be assessed by an isokinetic valve (PowerBreatheK5), using the best value obtained from 5 attempts, 'for this a continuous scale in cmH2O is used.
Muscle strenght of limbs | Baseline and then at the end of the 10-week training period.
  Ability of arm muscles to generate tension and overcome resistance. It is measured by the amount of force they can produce when pushing, pulling or lifting objects. This strength is essential for everyday activities such as walking, lifting, or playing sports. To assess the muscle function of lower limbs, we mesured through the Sit to Stand Test in 1 minute (STST-1m), with the values standardized for Chilean adults by Otto et al.
Muscle strenght of arms | Baseline and then at the end of the 10-week training period
  Ability of arm muscles to generate tension and overcome resistance. It is measured by the amount of force they can produce when pushing, pulling or lifting objects. This strength is essential for everyday activities such as walking, lifting, or playing sports. To assess the muscle function of arms, it will be evaluated by means of prehensile dynamometry, taking as reference values those established by Romero-Dapueto, et al. for Chilean adults.
Pulmonary Function | Baseline and then at the end of the 10-week training period
  Refers to the ability of the lungs to exchange oxygen and carbon dioxide between air and blood. It involves processes such as ventilation (air inflow and outflow), diffusion (passage of gases) and perfusion (pulmonary blood flow). For this study we will use the Forced Vital Capacity (FVC), the Forced Expiratory Volume in the first second (FEV1) measured in liters, and the ratio between both values (FEV1/FVC) established as a percentage. In addition, the statistical value obtained, according to the reference values of the Global Lung Function Initiative (GLI).
Treatment Adherence | Baseline and then at the end of the 10-week training period
  Extent to which a patient follows his or her physician's recommendations. It involves attending medical appointments and following lifestyle changes. Good adherence is crucial for successful treatment and improved health. Adherence will be measured in relation to the number of sessions the subject completes, i.e. completing the 20 training sessions counts as adherence and a lower number means non-adherence to treatment.
Adverse Effects | Baseline, in each of the training sessions and in the reevaluation.
  Unwanted reactions that may occur as a result of a treatment, such as the performance of a procedure. They can range from mild to severe. The American College of Sports Medicine has established a series of adverse effects of training, which we have listed and will be checked at each session to assess whether there were adverse effects of training. Among the problems that could occur are the following:
  1. Injuries
  2. Overload
  3. Dehydration
  4. Cardiovascular problems
  5. Gastrointestinal problems
  6. Neuroendocrine problems
  7. Others (to be noted manually by the trainer)
Functionality | Baseline and then at the end of the 10-week training period
  The ability of a system, object or person to perform the functions for which it was designed or adapted. It implies efficiency, utility and fitness for a specific purpose. In people, it refers to the ability to perform activities of daily living and participate in society. this parameter will be evaluated through the Activities of Daily Living Questionnaire (ADLQ-T).
Cognition | Baseline and then at the end of the 10-week training period
  Encompasses the mental processes that make it possible to acquire, process and use information. It includes functions such as attention, memory, language, perception, reasoning and problem solving. It is the basis of knowledge, learning and interaction with the environment. This parameter will be evaluated through the Montreal Cognitive Assessment (MoCA).

OTHER OUTCOMES:
Age | Baseline
  Number of years of age at study entry
Gender | Baseline
  Biological sex
Previous hospitalizations | Baseline
  Number of previous hospitalizations, since diagnosis
Years since diagnosis | Baseline
  Years since medical diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de La Frontera, Temuco, Cautín, Chile

IPD SHARING:
Plan to Share IPD: Yes
Study protocol
Supporting Information: Study Protocol
Time Frame: Five years since publication in Clinical Trials.
Access Criteria: All people, just contact for e-mail.
URL: https://postgrado.med.ufro.cl/index.php/investigacion

REFERENCES:
- See also: Web page of School of Medicine Universida de La Frontera — https://postgrado.med.ufro.cl/index.php/investigacion